CLINICAL TRIAL: NCT05198089
Title: The Development and Pilot of MyInSPO: an Individualized Spirituality Program for Oncology Patients to Improve Spiritual Well-Being
Brief Title: Development of a Digital Tool, MyInspiration, for the Improvement of Spiritual Well-Being in Patients with Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Timothy Pawlik, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: OSU-20390; NCI-2021-00630 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-12-20; First posted 2022-01-20 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Malignant Solid Neoplasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm I (MyInspiration) (Experimental): Patients use MyInspiration for spiritual and/or religious guidance for 30 days.
  Interventions: Other: Internet-Based Intervention

INTERVENTIONS:
Other: Internet-Based Intervention — Use MyInspiration website

SUMMARY:
The purpose of this study is to pilot a beta version of a digital resource that supports the religious and spiritual beliefs of cancer patients, "MyInspiration".After receiving a cancer diagnosis, survivors are encouraged to make major life-altering decisions related to their treatment and care. The availability of spiritual/religious resources during cancer treatment may positively impact patient outcomes, feelings of well-being, and be essential components of holistic, patient-centered care. MyInspiration is a digital tool focused on spiritual and/or religious guidance and support that can be customized based on patient preferences and administered to cancer patients and their family members during cancer treatment. MyInspiration may help improve spiritual well-being in patients with cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Conduct a pilot of MyInspiration to determine acceptability, feasibility, and general satisfaction by its end-users.

II. Explore the qualitative opinions of patients who participated in the feasibility trial more in-depth using 1-on-1 interviews.

OUTLINE: Single-group feasibility pilot.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Capacity to sign an informed consent form
* Eligible for a surgical procedure (defined with International Classification of Diseases [ICD]-10 codes) that will require an in-patient stay at the Ohio State University Comprehensive Cancer Center (OSUCCC)-James
* Diagnosed with cancer
* Ability to read English (however, we will make all possible considerations to include non-native English speakers)
* Access to some form of internet (webpage, smartphone, tablet, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Feasibility of MyInspiration:Recruitment | Up to 30 days
  Feasibility will be assessed by ratio of patients that enroll of the patients that indicate interest in the study
Feasibility of MyInspiration:Data Collection | Up to 30 days
  Feasibility will be assessed by completion rates of both the baseline and follow-up measures
Feasibility of MyInspiration:Usage Patterns | Up to 30 days
  Feasibility will be assessed by meta-analytics of website usage.
Acceptability of MyInspiration | Up to 30 days
  Acceptability will be assessed by study attrition rates.
General satisfaction of MyInspiration | Up to 30 days
  General Satisfaction will be assessed using an investigator-created 6-item scale assessing participants experience with MyInspo overall and its specific components

SECONDARY OUTCOMES:
Decisional regret | Up to 30 days
  Decisional regret will be assessed post cancer-directed surgery using The Decisional Regret Scale.Items will also be adapted from scales developed by Clark et al. regarding the perceptions of one's treatment decisions, their outcomes, and the inherent uncertainty of decision making and cancer control.
Spiritual well-being | Up to 30 days
  Spiritual well-being will be assessed using the Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being, the Meaning of Cancer Subscale from the Impact of Cancer scale, and 1-item assessing spiritual distress. The Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being is a 12-item scale with a minimum score of 0 and a maximum score of 48; higher scores indicate a greater sense of spiritual well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M Pawlik, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu